CLINICAL TRIAL: NCT02072265
Title: Utilization of a Medical Dual-spectrum Infrared Thermal Imaging System to Evaluate the Wound Healing of Permanently Implantable Venous Port (Port-A) and to Investigate the Relationship Between the Thermal Images and Subcutaneous/Bloodstream Infection
Brief Title: Using a Thermal Imaging System to Evaluate the Wound of Port-A and the Relationship Between Thermal Images and Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201309057RINC
Record Dates: First submitted 2014-02-12; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Wound Healing Disturbance of Port-A
Keywords: infrared thermal image; wound healing; wound infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Port-A implantation and chemotherapy: Patients scheduled for Port-A implantation and subsequent chemotherapy
  Interventions: Device: Infrared thermal images
- Port-A infection: Patients receiving Port-A removal due to infection
  Interventions: Device: Infrared thermal images

INTERVENTIONS:
Device: Infrared thermal images

SUMMARY:
Permanently implantable venous ports (Port-A) is very important to patients receiving chemotherapy. It not only provides a reliable route to administrate intravenous drugs, and it also requires minimal care when it is not in use. However, catheter related blood stream infection(CRBSI) is one of the serious complications of Port-A. The diagnosis of CRBSI relies on limited tools, including blood culture or symptoms and signs of active infection. In the stage of CRBSI, Port-A removal is necessary and pose the risk for the patients to re-implant the Port-A. Thus, it is crucial to early detect the infection and give appropriate treatment. Among the pathogens, some pathogens are related to skin contaminants. Before systemic spreading, these pathogens may colonize or cause minor infection subcutaneously. This investigation is to utilize a non-invasive dual spectrum infrared imaging system to evaluate the Port-A wound and to detect the infection.

Aim: 1. To build the database of infra-red thermal images of Port-A wound healing. 2. To investigate the thermal images of skin contamination related CRBSI and to compare with the thermal images of the CRBSI of unknown foci

ELIGIBILITY:
Inclusion Criteria:

* clinical requirement of chemotherapy with Port-A

Exclusion Criteria:

* not able to maintain posture during acquiring the thermal images
* with other wounds over the nearby area of the Port-A wound
* with other severe underlying disease and too weak to mobilize

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Port-A implantation and removal
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Port-A wound healing/infection status (infrared thermal images) | The patient will be followed once about 1 day before stitches removal of the port-A wound.
Port-A wound healing/infection status (infrared thermal images) | The patient will be followed once about 6 to 24 hours before the first chemotherapy
Port-A wound healing/infection status (infrared thermal images) | The patient will be followed once about 6 to 24 hours before the second chemotherapy
Port-A wound healing/infection status (infrared thermal images) | The patient will be followed once about 1 day before Port-A removal due to infection

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan